CLINICAL TRIAL: NCT07175298
Title: Efficacy of Serratus Posterior Superior Intercostal Plane Block on Post-operative Pain Management in Patients Undergoing Adult Cardiac Surgery. A Randomized Controlled Trial
Brief Title: Efficacy of Serratus Posterior Superior Intercostal Plane Block on Post-operative Pain in Cardiac Surgery.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Islam Elbardan, LECTURER OF ANESTHESIA AND SURGICALMINTENSIVE CARE, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0307518
Record Dates: First submitted 2025-09-15; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain; Cardiac Surgery
Keywords: The Serratus Posterior Superior Intercostal Plane Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: PCS fentanyl based (Active Comparator): Control Group: Participants will receive general anaesthesia with a conventional opioid-based technique(fentanyl)
  Interventions: Procedure: conventional opioid-based technique
- The Serratus Posterior Superior Intercostal Plane Block group (Experimental): SPSIPB Group: Participants will receive an ultrasound-guided Serratus posterior superior intercostal plane block with 30 ml 0.25% bupivacaine per side pre-incision and general anaesthesia with opioid based fentanyl
  Interventions: Procedure: SPSIPB Group

INTERVENTIONS:
Procedure: conventional opioid-based technique — Control Group: Participants will receive general anaesthesia with a conventional opioid-based technique
  Arms: Control Group: PCS fentanyl based
Procedure: SPSIPB Group — SPSIPB Group: Participants will receive an ultrasound-guided Serratus posterior superior intercostal plane block with 30 ml 0.25% bupivacaine per side pre-incision and general anaesthesia with opioid based fentanyl
  Arms: The Serratus Posterior Superior Intercostal Plane Block group

SUMMARY:
Cardiac surgery, particularly procedures involving median sternotomy, is associated with significant postoperative pain. Acute postoperative pain is severe in cardiac patients undergoing sternotomy, and pain intensity is more severe than expected. Poorly controlled pain after surgery can lead to myocardial ischemia and pulmonary infections.Regional anesthesia techniques offer a promising alternative or adjunct to systemic opioids, providing targeted pain relief with fewer systemic side effects. The Serratus Posterior Superior Intercostal Plane Block (SPSIPB) is a novel regional anesthesia technique that involves injecting local anesthetic into the fascial plane between the serratus posterior superior muscle and the intercostal muscles

DETAILED DESCRIPTION:
Cardiac surgery, particularly procedures involving median sternotomy, is associated with significant postoperative pain. Acute postoperative pain is severe in cardiac patients undergoing sternotomy, and pain intensity is more severe than expected. Poorly controlled pain after surgery can lead to myocardial ischemia and pulmonary infections.

Effective pain management is crucial for patient recovery, reducing complications, and facilitating early mobilization. Opioids are commonly used for postoperative analgesia but are associated with numerous side effects, including respiratory depression, nausea, vomiting, constipation, and prolonged hospitalization.

Regional anesthesia techniques offer a promising alternative or adjunct to systemic opioids, providing targeted pain relief with fewer systemic side effects. The Serratus Posterior Superior Intercostal Plane Block (SPSIPB) is a novel regional anesthesia technique that involves injecting local anesthetic into the fascial plane between the serratus posterior superior muscle and the intercostal muscles. This block will provide analgesia to the anterolateral and posterior chest wall, covering dermatomes relevant to cardiac surgery.

Preliminary case reports and small studies suggest its efficacy in thoracic and cardiac surgeries, demonstrating effective pain control and reduced opioid consumption. However, a randomized controlled trial is necessary to definitively determine the efficacy and safety of SPSIPB as part of multimodal analgesia in adult cardiac surgery.

Fascial plane blocks in regional anesthesia have gained importance in recent years. It involves injection into a tissue plane to provide analgesia and is an alternative to neuraxial and paravertebral techniques. It is often safer and is associated with less cardiorespiratory instability or complications compared to epidural analgesia.

The primary objective of the study is to examine the effect of adding preemptive SPSIPB to general anesthesia in adult cardiac surgery through sternotomy on the postoperative opioid consumption. The secondary objectives will include time to extubation, the intensity of postoperative pain, time to 1st rescue analgesia, patient satisfaction, and any possible side effects of the study drugs and technique.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 60
* both sexes
* who are scheduled to have fast-tracking elective on-pump cardiac surgery through a median sternotomy,
* American Society of Anesthesiologists Physical status II-III,
* Ability to understand and provide informed consent

Exclusion Criteria:

* patients who refused to participate in the study,
* who had Cognitive impairment or mental disorders,
* Ages <18 and >60 years,
* BMI <18 and >35,
* patients with puncture site infection,
* patients who documented allergy to local anesthetic drugs,
* patients used to take chronic pain medications, patients who made previous sternotomy or chest surgery
* patients with a history of substance abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Total postoperative fentanyl consumption | the first 24 and 48 hours post-extubation.
  will be measured as the total amount of fentanyl (in micrograms) consumed via PCA

SECONDARY OUTCOMES:
Time to extubation | post operative 6 hour
  duration (minutes) between ICU admission and endotracheal extubation.
Time to first rescue analgesia | 48hour post operatively
  Time from extubation to the first request for PCA bolus.
Postoperative pain intensity | 6, 12, 18,24, 36, and 48 hours post-extubation.
  Assessed using the Critical-Care Pain Observation Tool (CPOT) during intubation and the Numerical Rating Scale (NRS), at 6, 12, 18,24, 36, and 48 hours post-extubation. The CPOT ranges from 0 to 8, and the NRS ranges from 0 (no pain) to 10 (worst possible pain).
Patient satisfaction | at 24 hours post-extubation
  Assessed using a 5-point Likert scale ( 1-Very dissatisfied 2-Dissatisfied 3-Neutral 4-Satisfied 5-Very satisfied)
Length of stay | post operative 5 days
  total hospital stay (days).
Incidence of adverse | 28hour postoperative
  1. Related to local anesthesia toxicity (neurologic or cardiovascular events).
  2. Related to block procedure (hematoma and pneumothorax, nerve injury).
  3. Related to opioid administration (postoperative nausea and vomiting, dizziness, and pruritus, respiratory depression (respiratory rate < 10breaths/min or SpO2 < 90% on room air)).

CONTACTS AND LOCATIONS:
Overall Officials: Islam LECTURER OF ANESTHESIA AND SURGICAL INTENSIVE CARE, Dr, Principal Investigator — University of Alexandria
Locations (1):
- Faculty of medicine ,Alexandria university, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No